CLINICAL TRIAL: NCT03592199
Title: Biomarker Study of Patients With Metastatic Clear Cell Renal Carcinoma (ccRCC) Undergoing Sequential Therapy With 1st Line Sunitinib and 2nd Line Axitinib
Brief Title: Biomarker Study of Pts With Metastatic ccRCC Undergoing Sequential Therapy With 1st Line Sunitinib and 2nd Line Axitinib
Acronym: SuAx
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 1096/17
Record Dates: First submitted 2017-12-27; First posted 2018-07-19 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: biomarker; metastatic; sunitinib; axitinib; next generation sequencing; clear cell renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Sunitinib; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 1st Line Sunitinib and 2nd Line Axitinib (Experimental): 1st line sunitinib on a 4/2 schedule followed by axitinib 5 mg twice a day on 2nd line therapy
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — 1st line sunitinib on a 4/2 schedule followed by axitinib 5 mg twice a day on 2nd line therapy
  Other Names: Axitinib

SUMMARY:
This is a prospective single arm phase II study to evaluate potential prognostic and/or predictive biomarkers in patients with metastatic ccRCC undergoing treatment with 1st line sunitinib on a 4/2 schedule followed by axitinib on 2nd line therapy.

DETAILED DESCRIPTION:
In this study, all included patients will receive sunitinib until disease progression and/or limiting toxicity. If patients develop toxicities ≥ Grade 2 on 50 mg per day 4 weeks-on / 2 weeks-off schedule, a modified schedule of 50 mg/day 2 weeks-on / 1 week-off will be offered. After disease progression on sunitinib, all eligible patients will receive axitinib 5 mg twice a day. The investigators plan to assess, by next generation sequencing, the prevalence of mutations in several cancer related genes in baseline archived tissue from the patients included in the study, and the potential correlations between these somatic mutations and anti-VEGF (Vascular Endothelial Growth Factor) therapy efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Locally advanced (defined as disease not amenable to curative surgery or radiation therapy) or metastatic RCC (equivalent to Stage IV RCC according to American Joint Committee on Cancer staging) renal cell carcinoma;
* Histologic confirmed clear cell renal cell carcinoma;
* No prior systemic therapy (interleukin-2, interferon-α, chemotherapy, bevacizumab, sunitinib, sorafenib, pazopanib, axitinib, everolimus or temsirolimus) for advanced or metastatic RCC;
* Measurable disease by RECIST;
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2;
* Adequate organ system functions;
* Patients must understand and be willing to sign the written informed consent form of this study.

Exclusion Criteria:

* Non-clear cell renal cell carcinoma
* Pregnant or lactating female.
* History of another malignancy. Note: Subjects who have had another malignancy and have been disease-free for 3 years, or subjects with a history of completely resected non-melanoma skin carcinoma or successfully treated in situ carcinoma are eligible.
* History or clinical evidence of central nervous system (CNS) metastases. Note: Subjects who have previously-treated CNS metastases (surgery ± radiotherapy, radiosurgery) and meet all 3 of the following criteria are eligible:

  1. Are asymptomatic
  2. No evidence of active CNS metastases for ≥3 months prior to enrolment
  3. Have no requirement for steroids or anticonvulsants
* Clinically significant gastrointestinal abnormalities including, but not limited to:

  1. Malabsorption syndrome
  2. Major resection of the stomach or small bowel that could affect the absorption of study drug
  3. Active peptic ulcer disease
  4. Inflammatory bowel disease
  5. Ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation
  6. History of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within 28 days prior to beginning study treatment.
* History of any one or more of the following cardiovascular conditions within the past 12 months:

  1. Cardiac angioplasty or stenting
  2. Myocardial infarction
  3. Unstable angina
  4. Symptomatic peripheral vascular disease
  5. Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
  6. History of cerebrovascular accident including transient ischemic attack (TIA).
  7. Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥150 millimeters of mercury (mmHg) or diastolic blood pressure (DBP) of ≥ 90 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-12-11 (Estimated); Study Completion 2022-12-11 (Estimated)

PRIMARY OUTCOMES:
1st line Response Rate (RR) with Sunitinib in patients with VEGF pathway mutation | through study completion (up to 2 years)
  First Line Response Rate (RR) With Sunitinib (RECIST 1.1) in patients with VEGF pathway mutation

SECONDARY OUTCOMES:
1sr line RR with Sunitinib | through study completion (up to 2 years)
  First Line Response Rate (RR) with Sunitinib (RECIST 1.1)
2nd Line RR with Axitinib | through study completion (up to 2 years)
  Second Line Response Rate (RR) with Axitinib (RECIST 1.1)
1st line PFS with Sunitinib | through study completion (up to 2 years)
  First Line Progression Free Survival (PFS) with Sunitinib
2nd PFS with Axitinib | through study completion (up to 2 years)
  Second Line Progression Free Survival (PFS) with Axitinib
Overall Survival (OS) | through study completion (up to 2 years)
  Overall Survival
Incidence of Treatment-Emergent Adverse Events | through study completion (up to 2 years)
  CTCAE v.4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Cancer do Estado de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided